CLINICAL TRIAL: NCT02785315
Title: Cognitive Intervention for Persons With Amnestic Mild Cognitive Impairment: The Efficacy in Enhancement of Cognition and Complex Activities of Daily Living Function
Brief Title: Cognitive Intervention for Persons With Amnestic Mild Cognitive Impairment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 201402028RINC
Record Dates: First submitted 2016-05-18; First posted 2016-05-27 (Estimated); Last update posted 2019-03-14 (Actual); Status verified 2019-03

CONDITIONS: Mild Cognitive Impairment
MeSH Terms: conditions — Cognitive Dysfunction | interventions — Rehabilitation

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- rehabilitation & remediation approach (Experimental): The intervention group will receive 12 weekly 90-minute combined cognition interventions in a group. The first half of each session will be cognitive training which focus on teaching various cognitive strategies and their applications to enhance the attention, memory, processing speed, and executive functions. The second half of the session will apply rehabilitation intervention with various compensatory strategies. Investigators will use group discussion to discuss everyday situations with memory problem and specific strategies (internal and external) related to real-life situations. Investigators will also include one individual session in the 12 group sessions.
  Interventions: Behavioral: rehabilitation & remediation approach
- remediation approach (Active Comparator): The remediation approach will receive 12 weekly 90-minute cognitive training which focus on teaching various cognitive strategies and their applications to enhance the attention, memory, processing speed, and executive functions.
  Interventions: Behavioral: remediation approach

INTERVENTIONS:
Behavioral: rehabilitation & remediation approach — The rehabilitation & remediation approach group will receive 12 weekly 90-minute combined cognition interventions in a group. The first half of each session will be cognitive training which focus on teaching various cognitive strategies to enhance the attention, memory, processing speed, and executive functions. The second half of the session will apply rehabilitation intervention by discussing everyday situations with memory problem and specific strategies related to real-life situations. Investigators will also include one individual session in the 12 group sessions.
  Arms: rehabilitation & remediation approach
Behavioral: remediation approach — The remediation approach will receive 12 weekly 90-minute cognitive training which focus on teaching various cognitive strategies and their applications to enhance the attention, memory, processing speed, and executive functions.
  Arms: remediation approach

SUMMARY:
People with mild cognitive impairment (MCI) are at a greater risk of developing dementia. Therefore, it is important to develop effective non-pharmacological interventions to facilitate their cognitive and activities of daily living (ADL) function, which will also prevent or delay their progression to dementia and reduce associated healthcare and social costs. There are currently a variety of cognitive interventions, mainly categorized as remediation and rehabilitation approach. Research to compare their contents and effectiveness is strongly needed. The information can be used to individualize cognitive intervention based on specific cognitive profile of the patient.

This study aims to determine the immediate and long-term efficacy of the remediation approach and rehabilitation approach in enhancing the cognitive and ADL function. The research questions include 1) whether the rehabilitation approach compared with the remediation approach has better effects on improving ADL function; (2) whether the remediation approach may only enhance the performance on the cognitive tests rather than on the ADL function. This study will also explore whether the attitudes of caregivers on providing ADL assistance affect effects of cognitive intervention.

DETAILED DESCRIPTION:
The study is designed by a single-blinded randomized control trial. Sixty persons with MCI, confirmed by physicians, will receive 12 weekly 90-minute cognition interventions in a group of 6-8 persons. All participants will be randomly assigned to the following groups: 1) Remediation approach: various cognitive strategies will be taught, and exercises involving the practice of these strategies to enhance the attention, memory, processing speed, and executive functions. 2) Combination of rehabilitation and remediation approaches: The first half of each session will focus on the remediation approach as described above. The second half of the session will apply rehabilitation approach. The investigators will use group discussion to discuss everyday situations with memory problem and specific strategies (internal and external) related to real-life situations. The investigators will also include one individual session in the 12 group sessions.

All participants will be assessed at 3 time points: before intervention, right after intervention, and 12 weeks after the intervention. The primary outcomes are the ADL functions evaluated by subjective and objective measures, and cognitive function evaluated by tests of attention, memory and executive function. The secondary outcomes include the depression, the quality of life of the participants, and the caregivers' load. The intervention effects will be further analyzed by the caregivers' attitude regarding to the level of ADL assistance.

ELIGIBILITY:
Criteria: Inclusion Criteria:

* over 50 years old
* years of education > 6
* mild cognitive impairment diagnosed by physician
* no dementia diagnosis
* Barthel Index scored 100
* Geriatric Depression Scale-Short Form scored < 8

Exclusion Criteria:

* without concurrent major or significant psychiatric disorders
* severe physical diseases which might affect cognitive functions
* difficult to follow instructions due to visual or hearing impairments

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2014-12-16 (Actual); Primary Completion 2017-11-14 (Actual); Study Completion 2017-11-14 (Actual)

PRIMARY OUTCOMES:
Change from Baseline The Brief University of California San Diego (UCSD) Performance-Based Skills Assessment （Traditional Chinese Version）（UPSA-Brief ) at the 12th and 24th weeks | baseline, 12th and 24th weeks after intervention

SECONDARY OUTCOMES:
Change from Baseline Short-form Zarit Caregiver Burden Interview-12 (sCZBI-12) at the 12th and 24th weeks | baseline, 12th and 24th weeks after intervention
Change from Baseline Montreal Cognitive Assessment (MoCA) Taiwan Version at the 12th and 24th weeks | baseline, 12th and 24th weeks after intervention
Change from Baseline Word Sequence Learning Test at the 12th and 24th weeks | baseline, 12th and 24th weeks after intervention
Change from Baseline Minimal-Mental Status Exam (MMSE) at the 12th and 24th weeks | baseline, 12th and 24th weeks after intervention
Change from Baseline Miami Prospective Memory Test (MPMT) at the 12th and 24th weeks | baseline, 12th and 24th weeks after intervention
Change from Baseline Color Trails Test at the 12th and 24th weeks | baseline, 12th and 24th weeks after intervention
Change from Baseline Structure MRI at the 12th and 24th weeks | baseline, 12th and 24th weeks after intervention
Change from Baseline PiB-PET and FDG-PET at the 12th and 24th weeks | baseline, 12th and 24th weeks after intervention
  PiB-PET: Pittsburgh Compound B-Positron Emission Tomography FDG-PET:18-Fluoro-deoxyglucose positron emission tomography
Change from Baseline amyloid Aβ40, Aβ42 and tau proteins at the 12th and 24th weeks | baseline, 12th and 24th weeks after intervention
Change from Baseline The Disability Assessment for Dementia (DAD) at the 12th and 24th weeks | baseline, 12th and 24th weeks after intervention
Change from Baseline Quality of Life-Alzheimer's Disease scale (QoL-AD) at the 12th and 24th weeks | baseline, 12th and 24th weeks after intervention
Change from Baseline Goal Attainment Scaling (GAS) at the 12th and 24th weeks | baseline, 12th and 24th weeks after intervention
Change from Baseline Everyday Memory Questionnaire at the 12th and 24th weeks | baseline, 12th and 24th weeks after intervention

CONTACTS AND LOCATIONS:
Overall Officials: Hui-Fen Mao, Principal Investigator — National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No